CLINICAL TRIAL: NCT04043858
Title: Safety and Efficacy of Midodrine Hydrochloride in the Management of Refractory Ascites Due to Cirrhosis in Children: a Pilot Study
Brief Title: Safety and Efficacy of Midodrine Hydrochloride in the Management of Refractory Ascites Due to Cirrhosis in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Liver Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mid-Asci-Ped
Record Dates: First submitted 2019-08-01; First posted 2019-08-02 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Refractory Ascites; Children, Only
MeSH Terms: conditions — Ascites | interventions — Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Midodrine daily (Experimental): Midodrine hydrochloride 2.5 mg tab once per day
  Interventions: Drug: Midodrine 2.5 mg tab

INTERVENTIONS:
Drug: Midodrine 2.5 mg tab — Patients receive an oral daily dose of 2.5 mg midodrine if age 7-12 years and receive 2.5 mg twice daily of more than 12 years
  Other Names: ProAmatine

SUMMARY:
Ascites in liver cirrhosis is explained by increased production of vasoactive substances leading to renal vasoconstriction and salt and water retention. The retained water then accumulates in the peritoneal cavity under the effect of portal hypertension and low albumin. Refractory ascites is defined as ascites that cannot be mobilized or prevented from early recurrence after large-volume paracentesis despite medical therapy and dietary sodium restriction. Midodrine is an α1 receptor agonist that can improve systemic and renal hemodynamics in non-azotemic cirrhotic patients by counteracting mesenteric vasodilatation, which is accentuated in cirrhosis.

DETAILED DESCRIPTION:
Ascites in liver cirrhosis is explained by increased production of vasoactive substances, such as nitric oxide, carbon monoxide, and endocannabinoids, which cause splanchnic vasodilatation, increased blood flow through this area, and a decrease in peripheral vascular resistance and the effective arterial volume with resulting reduction in renal blood flow with subsequent activation of rennin-angiotensin-aldosterone system which in turn leads to renal vasoconstriction and salt and water retention. The retained water then accumulates in the peritoneal cavity under the effect of portal hypertension and low albumin.

The International Ascites Club defines refractory ascites as ascites that cannot be mobilized or prevented from early recurrence after large-volume paracentesis despite medical therapy and dietary sodium restriction.

There are two varieties of refractory ascites: diuretic-resistant ascites that is unresponsive to the maximal tolerable dose of diuretic therapy and diuretic-intractable ascites when complications such as hepatic encephalopathy, renal dysfunction, or electrolyte abnormalities limit the use of diuretics in the effective therapeutic dose (Cárdenas and Arroyo, 2005)

The therapeutic options for refractory ascites are serial therapeutic paracentesis, transjugular intrahepatic portosystemic shunt, peritoneovenous shunt, and liver transplantation.

Midodrine is transformed into the active metabolite desglymidodrine, which is an α1 receptor agonist causing an increase in vascular tone and increase in blood pressure without β-adrenergic receptors stimulation so, it can improve systemic and renal hemodynamics in non-azotemic cirrhotic patients by counteracting mesenteric vasodilatation, which is accentuated in cirrhosis. It diffuses poorly across the blood-brain barrier with no central effects.

In a study included 600 adult patients with refractory ascites, midodrine was added to diuretic therapy and lead to enhancement of diuresis with the improvement of systemic, renal hemodynamics and short-term survival. Approximately, the only use of midodrine hydrochloride in children was in postural orthostatic tachycardia syndrome (POTS) which showed a good efficacy and safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7-18 years
* Both sexes
* Having refractory ascites (not responding to maximal dose of diuretics
* Diuretic-induced complications necessitate discontinuation of the drug

Exclusion Criteria:

* Non-cirrhotic causes of ascites
* Intrinsic renal disease ( e.g; polycystic kidney disease)
* Active gastrointestinal bleeding or the presence of risky varices
* Patients with Portal vein thrombosis and Budd-Chiari
* Cardiovascular disease
* Systemic hypertension or prehypertension
* Hyperthyroidism
* Patients with narrow-angle glucoma

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-06-05 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Side effect no 1 | 3 months
  number of patients with Elevated BP: ≥90th percentile to <95th percentile
Side effect no 2 | 3 months
  number of patients with Stage 1 HTN: ≥95th percentile to <95th percentile + 12 mmHg or 130/80 to 139/89 mm Hg (whichever is lower)
Side effect no 3 | 3 months
  number of patients with Stage 2 HTN: ≥95th percentile + 12 mm Hg or ≥140/90 mm Hg (whichever is lower) mmHg or 130/80 to 139/89 mm Hg (whichever is lower)
Side effect no 4 | 3 months
  number of patients with low heart rate
Side effect no 5 | 3 months
  number of patients with urine retention
Side effect no 6 | 3 months
  number of patients with severe itching
Side effect no 7 | 3 months
  number of patients with skin rash

SECONDARY OUTCOMES:
Complete Response | 12 months
  absence of ascites by abdominal ultrasound
Partial response | 12 months
  ascites cannot be mobilized completely but not symptomatic or needs paracentesis
non-response | 3 months
  no decrease in ascites which still in need for paracentesis after 3 months of duration

CONTACTS AND LOCATIONS:
Overall Officials: Bassam Ayoub, MD, Principal Investigator — Pediatric Hepatology Dep; National Liver Institute, Menoufia University, Egypt
Locations (1):
- Pediatric Hepatology, Gastroenterology and Nutrition Department, National Liver Institute, Menoufia University, Shibīn al Kawm, Menofiya, Egypt

REFERENCES:
- [Background] Albillos A, Banares R, Gonzalez M, Catalina MV, Molinero LM. A meta-analysis of transjugular intrahepatic portosystemic shunt versus paracentesis for refractory ascites. J Hepatol. 2005 Dec;43(6):990-6. doi: 10.1016/j.jhep.2005.06.005. Epub 2005 Jul 5. PMID 16139922
- [Background] Bes DF, Cristina Fernandez M, Malla I, Repetto HA, Buamscha D, Lopez S, Martinitto R, Cuarterolo M, Alvarez F. Management of cirrhotic ascites in children: Review and recommendations. Part 2: Electrolyte disturbances, nonelectrolyte disturbances, therapeutic options. Arch Argent Pediatr. 2017 Oct 1;115(5):505-511. doi: 10.5546/aap.2017.eng.505. English, Spanish. PMID 28895701
- [Background] Cardenas A, Arroyo V. Refractory ascites. Dig Dis. 2005;23(1):30-8. doi: 10.1159/000084723. PMID 15920323
- [Background] Chen L, Wang L, Sun J, Qin J, Tang C, Jin H, Du J. Midodrine hydrochloride is effective in the treatment of children with postural orthostatic tachycardia syndrome. Circ J. 2011;75(4):927-31. doi: 10.1253/circj.cj-10-0514. Epub 2011 Feb 2. PMID 21301135
- [Background] Dionne JM. Updated Guideline May Improve the Recognition and Diagnosis of Hypertension in Children and Adolescents; Review of the 2017 AAP Blood Pressure Clinical Practice Guideline. Curr Hypertens Rep. 2017 Oct 16;19(10):84. doi: 10.1007/s11906-017-0780-8. PMID 29035421
- [Background] JCS Joint Working Group. Guidelines for drug therapy in pediatric patients with cardiovascular diseases (JCS 2012). Digest version. Circ J. 2014;78(2):507-33. doi: 10.1253/circj.cj-66-0083. Epub 2013 Dec 26. No abstract available. PMID 24369273
- [Background] Hanafy AS, Hassaneen AM. Rifaximin and midodrine improve clinical outcome in refractory ascites including renal function, weight loss, and short-term survival. Eur J Gastroenterol Hepatol. 2016 Dec;28(12):1455-1461. doi: 10.1097/MEG.0000000000000743. PMID 27622998
- [Background] Baker-Smith CM, Flinn SK, Flynn JT, Kaelber DC, Blowey D, Carroll AE, Daniels SR, de Ferranti SD, Dionne JM, Falkner B, Gidding SS, Goodwin C, Leu MG, Powers ME, Rea C, Samuels J, Simasek M, Thaker VV, Urbina EM; SUBCOMMITTEE ON SCREENING AND MANAGEMENT OF HIGH BP IN CHILDREN. Diagnosis, Evaluation, and Management of High Blood Pressure in Children and Adolescents. Pediatrics. 2018 Sep;142(3):e20182096. doi: 10.1542/peds.2018-2096. Epub 2018 Aug 20. PMID 30126937
- [Background] Moore KP, Wong F, Gines P, Bernardi M, Ochs A, Salerno F, Angeli P, Porayko M, Moreau R, Garcia-Tsao G, Jimenez W, Planas R, Arroyo V. The management of ascites in cirrhosis: report on the consensus conference of the International Ascites Club. Hepatology. 2003 Jul;38(1):258-66. doi: 10.1053/jhep.2003.50315. PMID 12830009
- [Background] Singh V, Dhungana SP, Singh B, Vijayverghia R, Nain CK, Sharma N, Bhalla A, Gupta PK. Midodrine in patients with cirrhosis and refractory or recurrent ascites: a randomized pilot study. J Hepatol. 2012 Feb;56(2):348-54. doi: 10.1016/j.jhep.2011.04.027. Epub 2011 Jul 13. PMID 21749847
- [Background] Tanaka H, Fujita Y, Takenaka Y, Kajiwara S, Masutani S, Ishizaki Y, Matsushima R, Shiokawa H, Shiota M, Ishitani N, Kajiura M, Honda K; Task Force of Clinical Guidelines for Child Orthostatic Dysregulation, Japanese Society of Psychosomatic Pediatrics. Japanese clinical guidelines for juvenile orthostatic dysregulation version 1. Pediatr Int. 2009 Feb;51(1):169-79. doi: 10.1111/j.1442-200X.2008.02783.x. PMID 19371306
- [Background] Zhang F, Li X, Ochs T, Chen L, Liao Y, Tang C, Jin H, Du J. Midregional pro-adrenomedullin as a predictor for therapeutic response to midodrine hydrochloride in children with postural orthostatic tachycardia syndrome. J Am Coll Cardiol. 2012 Jul 24;60(4):315-20. doi: 10.1016/j.jacc.2012.04.025. PMID 22813609